CLINICAL TRIAL: NCT02778178
Title: Analgesic Efficacy of Transversus Abdominis Plane (TAP) Block After Lumbar Spine Surgery Through Anterior Approach (Anterior Lumbar or Direct Lateral Interbody Fusion): a Prospective, Randomized, Double-blind Placebo-controlled Study
Brief Title: TAP Block Efficacy After Lumbar Spine Surgery Through Anterior Approach: a Randomized, Placebo-controlled Study
Acronym: TAP-LIF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-52; 2015-002143-34 (EudraCT Number)
Record Dates: First submitted 2016-05-18; First posted 2016-05-19 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Clonidine; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block with ropivacaine (Experimental): Bilateral single shot TAP block under ultrasound guidance: 20 mL ropivacaine 3.75 mg/ml + 75 µg clonidine, per side
  Interventions: Drug: ropivacaine plus clonidine; Device: ultrasound
- TAP block with placebo (Placebo Comparator): Placebo administration: bilateral single shot TAP block under ultrasound guidance: 20 mL saline 0.9%, per side
  Interventions: Drug: Placebo; Device: ultrasound

INTERVENTIONS:
Drug: ropivacaine plus clonidine — 20 mL ropivacaine 3.75 mg/ml + 75 µg clonidine, per side
  Arms: TAP block with ropivacaine
Drug: Placebo — 20 mL saline 0.9%, per side
  Arms: TAP block with placebo
Device: ultrasound

SUMMARY:
Anterior Lumbar Interbody Fusion (ALIF) as well as Direct Lateral Interbody Fusion (DLIF) are established techniques for lumbar interbody fusion. In contrast with posterior approaches, they allow free approach to the anterior disc space without opening of the spinal canal or the neural foramina. However, the additional anterior approach conveys specific concerns, including abdominal pain that may delay recovery after surgery. The transversus abdominis plane (TAP) block is a validated approach for postoperative pain relief following abdominal surgeries. There is currently no evidence of the possible benefits of TAP block as part of multimodal pain management after ALIF/DLIF surgery. The investigator hypothesize that a single-injection TAP block reduces opioid consumption after anterior lumbar fusion surgery. The main goal of this prospective, randomized, double-blind, placebo-controlled study is to demonstrate a >35% reduction in opioid consumption during the 24h following ALIF/DLIF surgery.

DETAILED DESCRIPTION:
Clinical trial : therapeutic, prospective, randomized,double blind, placebo-controlled, with parallel group, of superiority, in intention to treat, monocentric study.

The main steps of the study are:

* preoperative assessment of eligibility
* exclusion and inclusion criteria, written informed consent, baseline preoperative assessment (see specific section)
* randomization (using a computer generated list) immediately before induction of anesthesia
* TAP block: ropivacaine + clonidine (experimental group, n=20) OR saline (control group; n=20)
* anesthesia (propofol, sufentanil, cisatracurium, ketamine and desflurane) and postoperative analgesia (paracetamol, ketoprofen, nefopam, and patient-controlled analgesia with morphine) similar in both groups
* surgical procedure
* primary outcome parameter (morphine consumption first 24 hours; see specific section)
* secondary endpoints (see specific section, up to 6 months following surgery)

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over the age of 18 yr
* Patients with insurance coverage
* Patients able to provide free and informed consent
* Patients undergoing surgery by the ALIF or DLIF approaches

Exclusion Criteria:

* Patients receiving opioids as chronic treatment
* Patients with contra-indication to regional anesthesia or TAP block
* Patients unable to consent
* Patient refusal
* Patients with contra-indication to any drug included in the anesthesia or analgesia protocol
* Pregnancy or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | During the first 24 postoperative hours
  patient-controlled administration

SECONDARY OUTCOMES:
intraoperative sufentanil consumption | At the end of anesthesia
  infusion adjusted according to heart rate and arterial pressure
Sedation scale | During the first 6 hours
  using WHO Sedation scale
  - 0 = awake and alert /- 1 = quietly awake / - 2 = asleep but easily roused / - 3 = deep sleep
Morphine consumption | between the 24 and the 48 postoperative hours
  patient-controlled administration
Postoperative nausea and vomiting (PONV) Score | first 24 postoperative hours
  Measure the presence and severity of postoperative nausea and vomiting the PONV score :- 1 = mild /- 2 = moderate / - 3 = severe
Antiemetics consumption | During the first 24 postoperative hours
resumption of intestinal transit | Up to the end of hospital stay
visual analog scale | At Baseline, at wake up, during the first 48 postoperative hours, At 3 and 6 months after surgery
  Measure the pain severity
Area peri-incisional hyperalgesia | At 48 hours
  von frey's hair
Questionnaire Douleur de Saint-Antoine (QDSA) , | At Baseline, At 3 and 6 months after surgery
  evaluation with validated scores for chronic and neuropathic pains
Questionnaire d'Evaluation des Douleurs Neuropathiques (QEDN), | At Baseline, At 3 and 6 months after surgery
  evaluation with validated scores for chronic and neuropathic pains
Sullivan's "pain catastrophising scale", | At Baseline, At 3 and 6 months after surgery
  evaluation with validated scores for chronic and neuropathic pains
Hospital Anxiety and Depression Scale (HAD scale), | At Baseline, At 3 and 6 months after surgery
  evaluation with validated scores for chronic and neuropathic pains
Oswestry score | At Baseline, At 3 and 6 months after surgery
  evaluation with validated scores for chronic and neuropathic pains

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Tavernier, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Comite douleur-anesthesie locoregionale et le comite des referentiels de la Sfar. [Formalized recommendations of experts 2008. Management of postoperative pain in adults and children]. Ann Fr Anesth Reanim. 2008 Dec;27(12):1035-41. doi: 10.1016/j.annfar.2008.10.002. Epub 2008 Nov 21. No abstract available. French. PMID 19026514
- [Background] Tran TM, Ivanusic JJ, Hebbard P, Barrington MJ. Determination of spread of injectate after ultrasound-guided transversus abdominis plane block: a cadaveric study. Br J Anaesth. 2009 Jan;102(1):123-7. doi: 10.1093/bja/aen344. PMID 19059922
- [Background] Rozen WM, Tran TM, Ashton MW, Barrington MJ, Ivanusic JJ, Taylor GI. Refining the course of the thoracolumbar nerves: a new understanding of the innervation of the anterior abdominal wall. Clin Anat. 2008 May;21(4):325-33. doi: 10.1002/ca.20621. PMID 18428988
- [Background] Raoul S. Etude anatomique du nerf sinus vertébral. Thèse pour le Doctorat en Médecine. Faculté de Médecine de Lille (1996)
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] Belavy D, Cowlishaw PJ, Howes M, Phillips F. Ultrasound-guided transversus abdominis plane block for analgesia after Caesarean delivery. Br J Anaesth. 2009 Nov;103(5):726-30. doi: 10.1093/bja/aep235. Epub 2009 Aug 22. PMID 19700776
- [Background] Niraj G, Searle A, Mathews M, Misra V, Baban M, Kiani S, Wong M. Analgesic efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing open appendicectomy. Br J Anaesth. 2009 Oct;103(4):601-5. doi: 10.1093/bja/aep175. Epub 2009 Jun 26. PMID 19561014
- [Background] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789
- [Background] Farooq M, Carey M. A case of liver trauma with a blunt regional anesthesia needle while performing transversus abdominis plane block. Reg Anesth Pain Med. 2008 May-Jun;33(3):274-5. doi: 10.1016/j.rapm.2007.11.009. No abstract available. PMID 18433683
- [Background] Transversus Abdominal Plane Block. 52ème congrès national d'anesthésie et de réanimation. SFAR 2010